CLINICAL TRIAL: NCT05006482
Title: Optimizing Functional Outcomes of Older Cancer Survivors: The GEM-S Study
Brief Title: Geriatric Evaluation and Management With Survivorship Health Education for Older Survivors of Cancer, GEM-S Trial
Acronym: GEM-S
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Supriya Mohile, URCC Study Chair, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: URCC-19178; NCI-2021-01760 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC-19178 (Other: University of Rochester NCORP Research Base); URCC-19178 (Other: DCP); URCC-19178 (Other: CTEP); R01CA249467 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Malignant Solid Neoplasm
MeSH Terms: conditions — Lymphoma | interventions — Practice Guidelines as Topic; Standard of Care; Geriatric Assessment; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Survivors and caregivers receive routine survivorship follow-up care at their doctor's office for 3 visits over 6 months on study.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (GEMS intervention) (Experimental): Survivors and caregivers participate in GEMS consultation over 1 hour that includes discussion of results and recommendations from geriatric assessment. Both survivors and caregivers also participate in SHE sessions over 75 minutes twice weekly for 4 weeks. Survivors and caregivers also participate in EXCAP program, which includes daily walking and resistance exercises.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Educational Intervention; Other: Exercise Intervention; Other: Questionnaire Administration; Procedure: Tailored Intervention

INTERVENTIONS:
Other: Best Practice — Receive usual follow-up survivorship care
  Other Names: standard of care; standard therapy
  Arms: Arm I (usual care)
Other: Comprehensive Geriatric Assessment — Complete geriatric assessment
  Arms: Arm II (GEMS intervention)
Other: Educational Intervention — Participate in survivorship health education sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (GEMS intervention)
Other: Exercise Intervention — Participate in SHE-EXCAP program
  Arms: Arm II (GEMS intervention)
Other: Questionnaire Administration — Ancillary studies
Procedure: Tailored Intervention — Participate in GEM consultation
  Arms: Arm II (GEMS intervention)

SUMMARY:
This phase III trial compares the effect of geriatric evaluation and management with survivorship health education (GEM-S) to usual care on patient-reported physical function in older survivors of cancer. Survivorship care for older adults of cancer usually consists of getting advice from their doctor. This advice may include how to do their daily activities, so they are less tired or how to manage multiple diseases, or long-term side effects from treatment. GEM-S may help improve the physical ability to perform activities of daily living, mental well-being, and memory in older survivors of cancer after chemotherapy. This study may help doctors learn if including GEM-S in their practices improves physical, mental and memory functions in their patients. The study may also help to understand how such care affects cancer patients and their caregivers' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of GEM-S for improving patient-reported physical function (Functional Assessment of Chronic Illness-Fatigue Physical Well-Being Subscale [FACIT-PWB]) in older cancer survivors at 6 months. (Survivor Aim)

SECONDARY OBJECTIVE:

I. To assess the efficacy of GEM-S for improving patient-reported cognitive function (Functional Assessment of Cancer Therapy [FACT]-cognitive function [Cog]) in older cancer survivors at 6 months.

TERTIARY OBJECTIVES:

I. To assess the preliminary efficacy of GEM-S for improving:

Ia. Objective physical function (6-minute walk test) in older cancer survivors at 6 months; Ib. Objective cognitive function (Objective Cognitive Tests-Trail Making Part A/B [TMT A/B] and Controlled Oral Word Association [COWA] [i.e., FAS Test]) in older cancer survivors at 6 months.

EXPLORATORY HEALTH CARE OBJECTIVES:

I. To explore the preliminary efficacy of GEM-S for improving:

Ia. Survivor satisfaction with care (Health Care Climate Questionnaire [HCCQ] and communication about aging) at 6 months; Ib. Care coordination (# of contacts for co-management) up to 6 months; Ic. Survivor completion of referral appointments (# completed/# referrals) up to 6 months.

EXPLORATORY CAREGIVER OBJECTIVES:

I. To explore the preliminary efficacy of GEM-S for improving:

Ia. Caregiver distress (Distress Thermometer) at 6 months; Ib. Caregiver quality of life (Caregiver Quality of Life Index) at 6 months; Ic. Satisfaction with care (Health Care Climate Questionnaire [HCCQ] and communication about aging) at 6 months.

OUTLINE: Practice sites are randomized to 1 of 2 arms. Participants are assigned to arms based on practice site.

ARM I: Survivors and caregivers receive routine survivorship follow-up care at their doctor's office for 3 visits over 6 months on study.

ARM II: Survivors and caregivers participate in GEMS consultation over 1 hour that includes discussion of results and recommendations from geriatric assessment. Both survivors and caregivers also participate in survivorship health education (SHE) sessions over 75 minutes twice weekly for 4 weeks. Survivors and caregivers also participate in Exercise for Cancer Patients (EXCAP) program, which includes daily walking and resistance exercises.

After completion of study intervention, participants are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE CRITERIA: Participating practice clusters will be required to identify one (or more) oncologist and/or advanced practice practitioner (APPs; i.e., nurse practitioners, or physician assistants) as part of study eligibility. If another clinician is interested in participating, please contact University of Rochester Cancer Center (URCC) National Cancer Institute Community Oncology Research Program (NCORP) Research Base (RB) for approval

  * Oncologists/APPs/other clinicians must be licensed to practice
  * Oncologists/APPs/other clinicians must not have a plan to leave or retire from the NCORP practice within one year of enrolling into the study
* PRACTICE CRITERIA: Support/buy-in from oncology physicians and/or APPs and/or other clinicians who are willing to participate in training and study procedures and enroll cancer survivors
* ENTRY CRITERIA FOR ONCOLOGY PHYSICIANS/APPS/OTHER CLINICIANS: Oncology physicians/APPs/other clinicians must work at a participating site with no plans to leave that practice or retire within one year of enrollment into the study. We do not require that any or all oncology physicians and/or APPs at a practice setting agree to participate. Only one clinician is required for the practice cluster to be eligible. If another clinician (other than oncology physician or APP) is interested in participating, please contact URCC NCORP RB for approval
* CANCER SURVIVORS: 65 years or older
* CANCER SURVIVORS: Have completed or will have completed curative-intent treatment (e.g., surgery, chemotherapy, chemotherapy with radiation) for any solid tumor or lymphoma malignancy in last 6 months. If the survivor is receiving curative-intent chemotherapy, run-in study procedures can occur during the last 6 weeks of chemotherapy.

  * Cancer survivors who will receive or are receiving other treatments (e.g., hormonal treatment, monoclonal antibodies, immunotherapy, radiation) are eligible
  * For patients receiving neoadjuvant chemotherapy for curative intent, the run-in and baseline procedures can occur before or after surgery. Patients should be enrolled within 6 months from the end of surgery
* CANCER SURVIVORS: Be willing and able to come in for study visits or willing to undergo informed consent and assessments remotely via tele-health visits
* CANCER SURVIVORS: Be willing and able to provide informed consent and must sign consent in-person or remotely if it is not convenient or feasible to provide informed consent in-person
* CANCER SURVIVORS: Speak and understand English and/or Spanish. Spanish-speaking cancer survivors are eligible as long as there are appropriate resources in place for completion of study procedures at the practice site. Registration for Spanish-speaking cancer survivors must be approved by the URCC NCORP Research Base after a phone call to determine the feasibility for the practice to enroll a Spanish-speaking participant
* CAREGIVERS: 18 years or older
* CAREGIVERS: Selected by the cancer survivor when asked if there is a "family member, partner, friend or caregiver (age 18 years or older) with whom you discuss or who can be helpful in health-related matters." A caregiver need not be someone who lives with the cancer survivor or provides direct hands-on care
* CAREGIVERS: Speak and understand English and/or Spanish. Spanish-speaking caregivers are eligible as long as there are appropriate resources in place for completion of study procedures. Registration for Spanish-speaking caregivers must be approved by the URCC NCORP Research Base after a phone call to determine the feasibility for the practice to enroll a Spanish-speaking participant

Exclusion Criteria:

* CANCER SURVIVORS: Have a condition that precludes their ability to participate in informed consent or procedures (e.g., dementia)
* CAREGIVERS: Caregivers unable to understand the informed consent form or study procedures due to cognitive, health, or sensory impairment will be excluded

  * Capacity to conduct informed consent procedures and study procedures will be determined by the coordinators in collaboration with the cancer survivors' oncologists. These procedures are similar to that of URCC 13070, which enrolled caregivers of older patients with advanced cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Patient-reported physical function | Up to 6 months
  Will be assessed by the Functional Assessment of Cancer Therapy Physical Well-Being (FACIT-PWB) Subscale in older cancer survivors. The FACIT-PWB is 7-items as part of a larger 40-item FACIT-F questionnaire. Each question uses a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much).

SECONDARY OUTCOMES:
Patient-reported cognitive function | Up to 6 months
  Will be assessed by Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) Function in older cancer survivors. The FACT-Cog is a 37-item questionnaire, each with a 5-point Likert scale response. The FACT-Cog provides an overall score and subdomain scores (perceived cognitive impairment [PCI], perceived abilities, comments from others, and impact on quality of life). The secondary aim will be the PCI score at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Supriya G Mohile, Principal Investigator — University of Rochester NCORP Research Base
Locations (45):
- United States (45):
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Lake Regional Hospital, Osage Beach, Missouri
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Highland Hospital, Rochester, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Statesville, Stateville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - South Central Medical and Resource Center, Lindsay, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

REFERENCES:
- [Derived] Yilmaz S, Janelsins MC, Flannery M, Culakova E, Wells M, Lin PJ, Loh KP, Epstein R, Kamen C, Kleckner AS, Norton SA, Plumb S, Alberti S, Doyle K, Porto M, Weber M, Dukelow N, Magnuson A, Kehoe LA, Nightingale G, Jensen-Battaglia M, Mustian KM, Mohile SG. Protocol paper: Multi-site, cluster-randomized clinical trial for optimizing functional outcomes of older cancer survivors after chemotherapy. J Geriatr Oncol. 2022 Jul;13(6):892-903. doi: 10.1016/j.jgo.2022.03.001. Epub 2022 Mar 12. PMID 35292232